CLINICAL TRIAL: NCT05241912
Title: Supernormal Oxygen Delivery for Patients With Severe Burns：A Randomized Controlled Trial
Brief Title: Supernormal Oxygen Delivery for Patients With Severe Burns
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Liang Bing, Associate senior doctor, Guangzhou Red Cross Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-005-01
Record Dates: First submitted 2022-02-06; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Burn Surgery; Dobutamine
MeSH Terms: interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Intraoperative fluid management: administration of 6-10 ml/kg/hr of crystalloid solution.
- Goal-directed fluid group (Experimental): Intervention: administration of dobutamine 0.01 - 0.04 U/min after induction of anesthesia.
  Intraoperative fluid management: administration of 2-4 ml/kg/hr of crystalloid solution.
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — administration of dobutamine 0.01 - 0.04 U/min after induction of anesthesia to maintain oxygen delivery
  Arms: Goal-directed fluid group

SUMMARY:
This is a randomized double-blinded study to investigate in which the groups are designated as the control group and the goal-directed fluid therapy group to further evaluate significant differences in rate of complications during burn surgery.

DETAILED DESCRIPTION:
This is a randomized double-blinded study to investigate the effect of control group and the goal-directed fluid therapy group on complications during surgery of the burn patients. The groups are designated as the control group and the oal-directed fluid therapy group to further evaluate significant differences in complications during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Severe burn patients

Exclusion Criteria:

* Patients or families refuse to sign consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Complication | One week after operation
  perioperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Red cross hospital, Guangzhou, Guangdong, China